CLINICAL TRIAL: NCT02954289
Title: Increasing Healthy Outcomes for Prostate Cancer Survivors: An Innovative Cooking Class Intervention Pilot Study
Brief Title: Cooking Class Intervention Project for Men With Prostate Cancer and Their Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Carolyn Gotay, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 702413
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Prostate Cancer
Keywords: modifiable risk factors; lifestyle; nutrition; weight control; dietary intervention; health promotion; patient-partner outcomes; survivorship; prostate cancer outcomes
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary intervention (Other): Dietary intervention
  Interventions: Behavioral: Dietary intervention

INTERVENTIONS:
Behavioral: Dietary intervention — Session 1:The Breakfast Club: ways to increase the healthiness of breakfast and all meals.
  Session 2: Calcium and Vitamin D -Keys to Bone Health
  Session 3: Fruits and Veggies -Your New Best Friends
  Session 4: Let's Talk About Fat
  Session 5: Shopping Therapy
  Session 6: Celebrity Chefs Share Their Secrets
  Other Names: Cooking classes

SUMMARY:
Prostate cancer is one of the most commonly diagnosed cancers in Canada, with 24,000 new cases estimated for 2015. Prostate cancer patients often live with uncomfortable side effects of treatment, such as a decrease in bone health, weight gain, and challenges to their interpersonal relationships. Nutrition can improve outcomes for PCa survivors; however, dietary interventions for prostate cancer patients are limited. Therefore, this is a feasibility study that tests the impact of an innovative intervention to promote healthy nutrition and weight control for prostate cancer survivors and their partners.

The objectives are to assess the feasibility of the intervention, specifically:

* Accrual, retention and adherence, and participant satisfaction
* Candidate measures for primary outcomes in future studies

The intent is to evaluate how well the classes work and identify ways to make them more successful. At the end of the study, the investigators will know if this approach shows merit to be tested further through a randomized controlled trial.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most commonly-diagnosed invasive cancer in Canada, with 24,000 new cases predicted for 2015. The large majority of men (96%) will survive five or more years post-diagnosis. However, many PCa survivors live with side effects of the disease and treatment and may develop chronic conditions due to aging and/or cancer therapy. The PCa-related side effects can also impact men's interpersonal relationships. Effective interventions to promote health and well-being for PCa survivors are urgently needed.

Evidence shows that nutrition can improve outcomes for PCa survivors; however, dietary interventions for prostate cancer patients are limited. Furthermore, all PCa-related interventions reported thus far are limited in one important way: they focus only on the patient/survivor. Yet, the impact of prostate cancer extends to the spouse as well. When it comes to lifestyle interventions, responsibility for health behaviours and food preparation typically falls on the wife, particularly in today's cohort of PCa patients. As such, engaging the partner is crucial to ensure success for the survivor, and provide benefits for the wife as well.

Therefore, this is a feasibility study that tests the impact of an innovative intervention to promote healthy nutrition and weight control for PCa survivors and their partners.

The objectives are to assess the feasibility of the intervention, specifically:

* Accrual, retention and adherence, and participant satisfaction
* Candidate measures for primary outcomes in future studies

The study draws on Interdependence Theory and features of successful cooking class intervention research in other populations. Specifically, it uses hands-on cooking experience, combined with increased cooking skills and nutrition knowledge to build skills and self-efficacy; to be culturally appropriate and use simple affordable ingredients; and to involve the spouses.

The dietary intervention will be offered to a total of 24 couples (48 individuals). The intervention includes 6 cooking and nutrition-related classes, that are held weekly in a university classroom kitchen with interactive demo and cooking components. Classes focus on learning through preparing theme-based recipes, with themes organized around prostate health.

Feasibility outcomes are assessed throughout. Questionnaire-based outcomes are assessed pre- and post-intervention, anthropometric outcomes at first and last intervention session.

The main intent is to evaluate how well the classes work and identify ways to make them more successful. At the end of the study, the investigators will know if this approach shows merit to be tested further through a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria for Men with Prostate Cancer:

* A man
* Have a diagnosis of prostate cancer
* 18 years or older
* Are living with a wife or common-law partner
* Can read and understand English
* Have a desire to participate in a cooking class study with wife/partner

Exclusion Criteria for Men with Prostate Cancer:

• Are on a strict diet, such as gluten-free diet

Inclusion Criteria for Partners:

* Are a female
* Are living with a husband or common-law partner who has been diagnosed with prostate cancer
* Are 18 years or older
* Can read and understand English
* Have a desire to participate in a cooking class study with husband/partner

Exclusion Criteria for Partners:

• Are on a strict diet, such as gluten-free diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention as measured through study accrual | up to six weeks per session
Feasibility of the intervention as measured through participant adherence | up to six weeks per session
Feasibility of the intervention as measured through participant retention | up to 6 weeks per session
Feasibility of the intervention as measured through participant satisfaction interviews | 3-months post intervention

SECONDARY OUTCOMES:
Change in anthropometric measures (height, weight, hip and waist) | Baseline and 6 weeks
Change in relationship quality measured by the 15-item Mutuality Scale | Baseline and six weeks
Change in dietary outcome using a modified version of the National Institutes of Health Quick Food Scan | Baseline and 6 weeks
Change in quality of life using the 12-Item Short Form Health Survey | Baseline and six weeks
Change in quality of life using the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q) | Baseline and 6 weeks
Change in relationship using the Relationship Assessment Scale | Baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Gotay, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No